CLINICAL TRIAL: NCT05259436
Title: Collaborative Approach to Examining Adversity and Building Resilience Study
Acronym: CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Lifelong Medical Care (Unknown); UCSF Benioff Children's Hospital Oakland (Other); Santa Barbara Neighborhood Clinics (Unknown); University of California, Santa Barbara (Other); Futures Without Violence (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-34534
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Early Life Adversity; Caregiver Stress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Wait-list randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to the caregiver-child intervention using a block allocation scheme. Given the nature of the intervention the participants and their healthcare providers will be unblinded to their assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver-Child Intervention (Experimental): Investigators will examine the immediate psychosocial, behavioral, and child biologic response to three caregiver-child interventions depending on site of enrollment. Each interventions contain overlapping core elements, but also contribute unique facets, allowing us to examine overall intervention effects, as well as unique settings (e.g. home vs. clinic) and delivery effects (1:1 vs. group), providing insight for future direction.
  Interventions: Behavioral: Caregiver-child Intervention
- Enhanced Primary Care (Active Comparator): Navigational services for social need resources.
  Interventions: Behavioral: Enhanced Primary Care

INTERVENTIONS:
Behavioral: Caregiver-child Intervention — Intervention Groups:
  1. Resilience Clinic (Benioff Oakland): 6 weekly interactive group-based visits in primary care that draws from the evidence-based Circle of Security Parenting along with the principles of mindfulness;
  2. ABC Intervention (Lifelong): 10 weekly home visiting sessions. ABC is an empirically supported parenting program that focuses on improving maternal sensitivity;
     and,
  3. Resiliency Family Program (Santa Barbara Neighborhood Clinic): 4 primary-care-based visits, every 2-3 weeks, that include psycho-education materials drawing from the culturally-responsive, evidence-based program, Madres a Madres.
  Arms: Caregiver-Child Intervention
Behavioral: Enhanced Primary Care — Enhanced Primary Care (control group): This includes care coordination services for community resources in addition to usual care. Participants will be asked about any unmet social needs, e.g. food insecurity, financial strain, safe places to play. Those who endorse need will be offered navigational services to link to community resources.
  Arms: Enhanced Primary Care

SUMMARY:
To examine the behavioral, psychosocial, and biologic impact of resilience-promoting interventions associated with primary care.

DETAILED DESCRIPTION:
Early-life trauma and related adversities are prevalent and associated with negative health and achievement outcomes. These adverse childhood experiences (ACEs) are especially common in economically disadvantaged and communities of color. While there has been tremendous growth in knowledge about ACEs and their impact on health across the life course, critical gaps persist: 1) Which biologic pathways are most affected by ACEs during early childhood and may help identify those children at greatest risk for future poor health? And, 2) How may child and family resilience be bolstered across the care continuum to mitigate the negative health effects of ACEs? These critical gaps severely limit our ability to effectively identify children at high-risk and to intervene to promote resilience before poor health occurs.

Three previously piloted resilience-promoting, caregiver-child interventions will be examined: primary care-based, group-delivered Resilience Clinic (RC); home-based, dyadic Attachment and Biobehavioral Catch-up (ABC); and primary care-based, dyadic Resiliency Family Program (RFP). Using a randomized wait- list controlled trial design,12 families will be assigned to intervention or enhanced primary care (n=50/arm in each intervention, total n=300). Pre-post intervention health (behavioral, caregiver stress) and biology will be compared between intervention and controls, as well as modifying factors such as setting and delivery method.

ELIGIBILITY:
Inclusion Criteria:

1. Regular access to web-based computer, smart phone, or tablet if necessary to delivery via telehealth due to the COVID19 Pandemic (relative exclusion criteria - have budgeted to provide tablets and mobile wifi hot spots for up to 10% of participants)
2. Attachment and Biobehavioral Catch-up (ABC) Program

   * Caregiver: 18 years old and older, primary caregiver, English or Spanish speaking
   * Child: 2 to 4 years, PEARLS score > 1
3. Resilience Clinic

   * Caregiver: 18 years old and older, primary caregiver, English or Spanish speaking
   * Child: 2 to 5 years, PEARLS score > 1 or verbal disclosure of PEARLS adversity to primary care clinician/staff
4. HEROES Family Program

   * Caregiver: 18 years old and older, primary caregiver, ACE score > 2 if child PEARLS score = 0, English or Spanish speaking
   * Child: 2 to 5 years, PEARLS score > 1

Exclusion Criteria:

1. Caregiver: active suicidality, other psychiatric issues
2. Child: significant medical co-morbidities (i.e. disease requiring immunomodulators, chemo or radiation therapy, or hormonal therapy)

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Parenting Stress Index (PSI) score | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  Caregiver reported survey validated measure of parenting stress. The Parenting Stress Index - Short Form (PSI) is a 36-item self-report measure completed by parents to measure stress level within the context of parenting. Participants respond to items on a 5-point Likert scale. Responses to each item in a sub-category are totaled to calculate three subcategory scores, which are summed to represent a total parenting stress score. Higher scores indicate higher levels of parenting stress.
Change in Child Behavior Checklist (CBCL) total problems scale score | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  Caregiver reported survey validated measure of child behavioral and emotional challenges on the Child Behavior Checklist (CBCL) Preschool form from The Achenbach System of Empirically Based Assessment (ASEBA). The CBCL is standardized for children ages 1.5 to 5 years. Respondents are asked to rate 99 problem items as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child" based on the past two months. The range of possible values is 0-100.

SECONDARY OUTCOMES:
Change in global health (PROMIS global health) | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  PROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. This study uses the first question on the global scale, with minimum value of 1 and maximum of 5. Higher scores mean better general health.
Change in caregiver depression (PHQ) total score | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  Caregiver reported survey validated measure of self-report depressive symptoms on the Patient Health Questionnaire (PHQ). Respondents are asked 8 questions to rate from 0 for "not at all" to 3 for "nearly every day" based on the past two weeks. The range of possible values is from 0-27. Higher scores indicate higher self-report depressive symptoms.
Change in caregiver anxiety (GAD) total score | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  Caregiver reported survey validated measure of self-report symptoms of general anxiety on the General Anxiety Disorder (GAD) questionnaire. Respondents are asked 7 questions to rate from 0 for "not at all" to 3 for "nearly every day" based on the past two weeks. The range of possible values is from 0-21. Higher score indicates higher self-report general anxiety symptoms.
Change in family cohesion total score | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  The Family Adaptability and Cohesion Evaluation Scales II (FACES II) family cohesion scale evaluates eight concepts (2 items each): emotional bonding, family boundaries, coalitions, time, space, friends, decision-making, and interest and recreation. Respondents rate from 1 for "almost never or never" to 5 for "almost always or always." A higher score indicates high family cohesion.
Change in adult reported social and emotional support (ARSES) total score | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  Adult-reported social and emotional support is assessed using a standardized single item, "How often do you get the social and emotional support you need?" Response choices were "always," "usually," "sometimes," "rarely," or "never."
Change in atopy (ISSAC screen) | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  ISAAC was an epidemiological study following a survey of 2 million children worldwide to evaluate the prevalence of atopic disease in various ethnic backgrounds. The questionnaire is self-reported by parents and children to evaluate asthma, allergic rhinitis and eczema in childhood. 21 items, core questionnaires to assess the prevalence and severity of asthma, rhinitis and eczema in defined populations.
Change in general stress (Perceived Stress Scale) total score | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  The Perceived Stress Scale measures the extent to which an individual perceives situations in his or her life as stressful. It is a measure of global perceived stress and asks about feelings and thoughts during the last month. Respondents are asked 10 questions to rate from 0 for "never" to 4 for "very often" based on the past month. The range of possible values is from 0-40. Higher score indicates higher perceived stress.
Change in health-related social needs (Accountable Health Communities total score) | baseline/enrollment and 2 week and 3-month follow-up after intervention ends
  Questionnaire assessing impacts of current unmet health-related social needs (6 items; housing instability and problems, food insecurity, transportation needs, problems paying for utilities/bills) and number of current social needs.
  Questionnaire assessing impacts of current unmet health-related social needs (6 items; housing instability and problems, food insecurity, transportation needs, problems paying for utilities/bills) and number of current social needs.
  Questionnaire assessing impacts of current unmet health-related social needs (6 items; housing instability and problems, food insecurity, transportation needs, problems paying for utilities/bills) and number of current social needs.
Telomere length | baseline/enrollment and 3-month follow-up after intervention ends
  Telomeres are nucleoproteins that protect the ends of chromosomes. Telomere length is a biomarker of cellular aging. Chronic stress has been associated with shorter telomere length.
Leptin | baseline/enrollment and 3-month follow-up after intervention ends
  Leptin is a hormone primarily secreted by fat cells to reduce hunger.
CRP | baseline/enrollment and 3-month follow-up after intervention ends
  C-reactive protein is produced by the liver in response to inflammation. Higher level of CRP in the blood is an indicator of inflammation.
IGFBP1 | baseline/enrollment and 3-month follow-up after intervention ends
  Insulin-like growth factor binding protein 1 is mainly expressed in the liver and circulates in plasma where it interacts with IGF-1 and 2. IGFBP-1 plays an important role in metabolism and low levels of this protein has associated with impaired glucose tolerance and hypertension
HA1C | baseline/enrollment and 3-month follow-up after intervention ends
  The hemoglobin A1c (glycated hemoglobin, glycosylated hemoglobin, HbA1c, or A1c) test is used to evaluate a person's level of glucose control. The test shows an average of the blood sugar level over the past 90 days and represents a percentage.
blood pressure | baseline/enrollment and 3-month follow-up after intervention ends
  Systolic and diastolic blood pressure, averaged across 3 readings.
resting heart rate | baseline/enrollment and 3-month follow-up after intervention ends
  Number of beats per minutes.
waist circumference | baseline/enrollment and 3-month follow-up after intervention ends
  Measuring waist circumference in cm. Waist and hip measurements will be combined to report waist-hip ratio (WHR) as a dimensionless ratio of the circumference of the waist to that of the hips.
hip circumference | baseline/enrollment and 3-month follow-up after intervention ends
  Measuring hip circumference in cm. Waist and hip measurements will be combined to report waist-hip ratio (WHR) as a dimensionless ratio of the circumference of the waist to that of the hips.
weight | baseline/enrollment and 3-month follow-up after intervention ends
  Weight will be measured in kg. Weight and height will be combined to report BMI in kg/m^2
height | baseline/enrollment and 3-month follow-up after intervention ends
  Height will be measured in cm. Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Thakur, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - LifeLong Medical Care, Richmond, California
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - Santa Barbara Neighborhood Clinics, Santa Barbara, California

IPD SHARING:
Plan to Share IPD: No